CLINICAL TRIAL: NCT00047203
Title: A Phase II Study of Flavopiridol in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: Flavopiridol in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02496; MC018B; N01CM17104 (NIH); CDR0000257567 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — alvocidib

ARMS (1):
- Treatment (flavopiridol) (Experimental): Patients receive flavopiridol IV over 1 hour on days 1-3. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients achieving at least a partial response may continue treatment in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275

SUMMARY:
Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Phase II trial to study the effectiveness of flavopiridol in treating patients who have relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with relapsed or refractory multiple myeloma treated with flavopiridol.

II. Determine the disease-free survival and overall survival of patients treated with this drug.

III. Correlate disease response with t(11;14)(q13;q32) rearrangement, p16 methylation status, and BCRP expression in patients treated with this drug.

IV. Correlate disease response and drug treatment with cell cycle status and effects on apoptosis and apoptosis regulatory proteins in these patients.

OUTLINE: This is a multicenter study.

Patients receive flavopiridol IV over 1 hour on days 1-3. Courses repeat every 21 days for up to 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients achieving at least a partial response may continue treatment in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory multiple myeloma (MM) requiring treatment

  * Durie-Salmon stage I or greater at diagnosis

    * Patients with non-secretory or oligo-secretory MM (defined as maximum urinary M-spike less than 200 mg/24 hours and a maximum serum M-spike less than 0.5 g/dL during entire disease course) must have at least 30% bone marrow plasma cells
    * Patients with secretory MM must have measurable disease defined as serum monoclonal protein of at least 1 g/dL or urinary M-spike of at least 200 mg/24 hours
* Must have received at least 1, but no more than 5 prior therapy regimens

  * Patients who have had 4 or 5 regimens are allowed provided corticosteroids and/or thalidomide are part of the regimens
  * No more than 5 prior chemotherapy regimens (as long as 2 contained dexamethasone or thalidomide)
  * Prior autologous peripheral blood stem cell transplantation is considered 1 prior regimen
* Performance status - ECOG 0-2
* Performance status - ECOG 0-3 if secondary to neuropathy or acute bone event (e.g., vertebral compression or rib fracture)
* Absolute neutrophil count at least 750/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN
* AST no greater than 2.5 times ULN
* Creatinine no greater than 3 mg/dL
* No myocardial infarction within the past 6 months
* Peripheral neuropathy secondary to prior drug therapy or myeloma-associated neuropathy allowed
* No other uncontrolled serious medical condition
* No uncontrolled infection
* No other active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* No prior allogeneic stem cell transplantation
* At least 10 days since prior thalidomide
* No concurrent biologic therapy
* See Disease Characteristics
* At least 2 weeks since prior myelosuppressive chemotherapy
* No other concurrent chemotherapy
* See Disease Characteristics
* No concurrent corticosteroids (including as antiemetics) except chronic corticosteroids for disorders other than myeloma (e.g., rheumatoid arthritis or adrenal insufficiency)

  * Maximum dose allowed for prednisone is no more than 10 mg/day or hydrocortisone no more than 40 mg/day
* At least 10 days since prior bortezomib or tipifarnib
* Concurrent bisphosphonates allowed if on stable dose before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-09; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Confirmed response (CR, VGPR, or PR) defined as a patient who has achieved response and maintained it on two consecutive evaluations at least 4 weeks apart. | First 3 months of treatment
  Ninety percent confidence intervals for the true success proportion will be calculated assuming a binomial distribution.

SECONDARY OUTCOMES:
Overall survival time | Time from registration to death due to any cause, assessed up to 1 year
  The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time to disease progression | Time from registration to documentation of disease progression, assessed up to 1 year
  The distribution of time to progression will be estimated using the method of Kaplan-Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States